CLINICAL TRIAL: NCT07017855
Title: Stereotactic Radiosurgery as Second-line Therapy for Ventricular Tachycardia
Acronym: STAR-4VT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/ABM/01/00031
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Ventricular Tachycardia, Monomorphic; Ventricular Tachycardia, Sustained; Ventricular Tachycardia (VT); Ventricular Tachycardia (V-Tach); Stereotactic Body Radiation Therapy (SBRT); Stereotactic Techniques; Stereotactic Radiation; Cardioverter-Defibrillators, Implantable
Keywords: Ventricular Tachycardia; VT; Stereotactic Arrhythmia Radioablation; STAR; Implanted Cardioverter-Defibrillator; ICD
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Eligible consecutive patients who provide written informed consent will be randomly assigned to one of two groups: (1) an experimental group in which patients will undergo the STAR procedure (radioablation) and (2) a control group in which patients will undergo standard endocardial catheter ablation (electrophysiology) using radiofrequency current. The allocation ratio for both groups will be 1:1.
  A stratified randomization method with block randomization will be applied using a centralized randomization system. The stratification factors will include sex and left ventricular ejection fraction (LVEF) (≤40% vs. >40%). Each participant will be assigned to one of the study arms, and follow-up will be conducted in a parallel study design. Due to the distinct nature of the interventional procedures, blinding of the study will not be feasible.
Masking Description: Due to the distinct nature of the interventional procedures, blinding of the study is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stereotactic Arrhythmia Radioablation (STAR) procedure (Experimental): In the arm randomized to STAR (alternative experimental therapy), the procedure will involve the elimination of the sVT substrate using ionizing radiation at a dose of 25 Gy, employing highly conformal stereotactic techniques. The STAR procedure will be performed in a radiation oncology department according to a protocol developed by the research team, based on the American Association of Physicists in Medicine (AAPM) report on stereotactic radiotherapy, guidelines for radiotherapy in patients with cardiac implantable electronic devices (CIEDs), and the expert consensus on the implementation and use of STAR in treatment-resistant sVT.
  Interventions: Radiation: Stereotactic Arrhythmia Radioablation (STAR)
- Active Comparator: Catheter Ablation using Radiofrequency Current (Active Comparator): In the arm randomized to CA (reference - standard therapy), the procedure will involve the elimination of the sVT substrate using energy transmitted from a generator through a catheter. The CA procedure will be performed in accordance with the expert consensus of the Heart Rhythm Society (HRS), European Heart Rhythm Association (EHRA), Asia Pacific Heart Rhythm Society (APHRS), and Latin American Heart Rhythm Society (LAHRS) on ventricular arrhythmia ablation.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Radiation: Stereotactic Arrhythmia Radioablation (STAR) — Radiotherapy Implementation: During treatment on a TrueBeam™ linear accelerator (Varian Medical Systems, Palo Alto, CA, USA), a planned radiation dose of 25 Gy will be delivered to the defined planning target volume (PTV) using highly conformal stereotactic techniques. Image-guided radiotherapy (IGRT), respiratory gating, and Triggered Tracking will be utilized, targeting the previously delineated defibrillation lead of the implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D), with position verification every 15 degrees of gantry rotation.
  Patient positioning will be performed using kV-kV imaging, based on pre-determined fiducial markers on the ICD/CRT-D defibrillation lead, followed by verification using gated cone-beam computed tomography (CBCT). Continuous ECG monitoring will be conducted throughout the treatment, and the patient will remain under cardiologist supervision.
  Arms: Stereotactic Arrhythmia Radioablation (STAR) procedure
Procedure: Catheter Ablation — CA will be conducted in an electrophysiology laboratory and will routinely follow diagnostic procedures, including an electrophysiological study (EPS) and three-dimensional electroanatomical mapping (3D-EAM). Once sufficient data on the nature and location of the arrhythmic substrate have been obtained from the three primary mapping modules-voltage, activation, and propagation-spatial 3D-EAM maps will be integrated with a 3D left ventricular reconstruction from multislice computed tomography (MSCT) or cardiac magnetic resonance (CMR). Subsequently, ablation will be performed by delivering energy to predefined target sites identified as the arrhythmia source to close the sVT isthmus or eliminate late potentials (LPs) and/or low-amplitude ventricular activities (LAVAs). Following CA, a repeat induction attempt of sVT using programmed ventricular pacing (VP) will be conducted to verify procedural efficacy.
  Arms: Active Comparator: Catheter Ablation using Radiofrequency Current

SUMMARY:
The aim of the study is to compare the efficacy and safety of treating recurrent sustained Ventricular Tachycardia (sVT) after prior Catheter Ablation (CA) in patients with Implanted Cardioverter-Defibrillator (ICD) between re-do of conventional endocardial CA and Stereotactic Arrhythmia Radioablation (STAR).

DETAILED DESCRIPTION:
Study Objectives:

To evaluate the safety and efficacy of Stereotactic Arrhythmia Radioablation (STAR) as a second-line therapy for sustained Ventricular Tachycardia (sVT) in optimally treated patients following endocardial Catheter Ablation (CA).

Study Design:

This study is a single-center randomized, noninferiority, head-to-head control trial comparing the efficacy and safety of two ablation methods for recurrent sVT after failing CA.

Patient Population:

Optimally treated patients aged ≥18 with Implantable Cardioverter-Defibrillators (ICD) in the primary or secondary prevention of sudden cardiac death (SCD), who have undergone endocardial CA and are candidates for re-ablation of recurrent symptomatic ventricular tachycardia (VT) following the 2022 European Society of Cardiology Guidelines for the management of patients with ventricular arrhythmias and the prevention of SCD.

The planned size of the group is 150.

The planned recruitment period is 42 months, and the observation period is 18 months.

Patients will be randomly assigned to experimental and control groups for a 1:1 group size ratio. The block randomized stratification method will be used with a central randomization system. Sex and left ventricular ejection fraction (≤40% vs. >40%) will be stratifying factors.

Intervention:

The intervention under investigation (experimental) will be STAR ablation. The standard intervention will be repeated endocardial radiofrequency CA. The target area for sVT ablation will be the arrhythmogenic substrate, defined by electrophysiological study (EPS) with three-dimensional electroanatomical mapping (obligatory in the standard therapy arm, optional in the STAR arm) and imaging tests (i.e., MSCT/CMR/PET-CT). The following will be integrated using dedicated computer software: 1) anatomical data-locating the arrhythmogenic scar area with channels of heterogeneous tissue-obtained using MSCT, CMR, PET-CT/SPECT, 2) three-dimensional electroanatomical maps-locating electrograms showing low peak-to-peak voltage, local abnormal ventricular activities, the sequence of myocardial activation, and critical isthmus sites for re-entrant VT, and 3) electrocardiograms detected during sinus rhythm and ventricular pacing during EPS. In the experimental arm, the obtained data will become the basis for STAR planning by a team consisting of a diagnostic cardiologist, radiologist, electrophysiologist, and radiotherapist. The obtained data will become the basis for endocardial CA planning in the control arm.

Observation:

Observation will include 1) clinical assessment-with the determination of the New York Heart Association functional class and exercise capacity in the 6-minute walk test (6MWT); 2) echocardiography-with the assessment of global and segmental left ventricular systolic function, mitral valve function, and the presence of fluid in the pleural and pericardial cavities; 3) parameters of pacing, sensing, lead impedance, and ventricular arrhythmic events recorded by the ICD/CRT-D; 4) QoL; and 5) procedure-related adverse events. Evaluation will be performed at 1, 3, 6, 12, and 18 months post-procedure, with endpoints assessed at 6 and 18 months.

The co-primary endpoints will assess 1) treatment efficacy, defined as the number of events of monomorphic sVT over six months following the comparison procedures, and 2) treatment safety, defined as no procedure-related serious adverse events.

The most important clinical parameters evaluating the effectiveness of ablation (i.e., post-procedural reduction in the sVT burden, occurrence/time to the first sVT episode, number of adequate ICD/CRT-D therapies, number of hospitalizations for arrhythmic reasons, QoL improvement) and mortality (death from any cause) were selected as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of enrollment.
2. Presence of structural heart disease (SHD) of either ischemic or non-ischemic etiology.
3. Implanted ICD or CRT-D device for primary or secondary prevention of sudden cardiac death (SCD).
4. History of at least one endocardial CA procedure targeting a substrate of monomorphic sVT.
5. Recurrence of at least one clinically significant and symptomatic episode of monomorphic sVT.
6. Optimal pharmacological treatment of underlying SHD, including maximally tolerated doses of guideline-recommended heart failure therapies and appropriate antiarrhythmic management.
7. Provision of written informed consent prior to study participation.

Exclusion Criteria:

1. Reversible cause of sVT recurrence, particularly acute coronary syndrome (ACS), acute myocarditis, or lead-related infective endocarditis (LDIE).
2. Myocardial infarction (MI) or cardiac surgery within the last 40 days.
3. Idiopathic sVT unrelated to SHD or sVT associated with genetically determined channelopathies.
4. Ongoing or persistently recurrent hemodynamically unstable sVT until clinical stabilization is achieved.
5. Acute decompensation of heart failure, classified as New York Heart Association (NYHA) Class IV, until clinical stabilization is achieved.
6. Worsening angina, classified as Canadian Cardiovascular Society (CCS) Class III or IV until coronary diagnostic evaluation and clinical stabilization are completed.
7. A mobile thrombus within the left ventricle (LV).
8. Presence of a left ventricular assist device (LVAD).
9. Presence of comorbidities or known risk factors for CA complications that, in the judgment of the electrophysiologist, constitute a contraindication to the procedure for safety reasons.
10. Active, uncontrolled malignancy and/or chemotherapy or immunotherapy administered or planned within 1 month of the scheduled ablation procedure.
11. Features of an active systemic, pulmonary, or pericardial inflammatory process requiring systemic treatment (disease-modifying therapies, corticosteroids, immunosuppressants) within the past 6 months.
12. Presence of comorbidities or known risk factors for radiotherapy complications that, in the judgment of the radiation oncologist, constitute a contraindication to STAR for safety reasons.
13. Pregnancy or breastfeeding.
14. Systemic disease that limits the probability of survival to less than 1 year
15. Other comorbidities, addictions, or social indications that, in the investigator's opinion, would preclude practical cooperation or otherwise disqualify the patient from participation in the clinical study.
16. Refusal to participate or lack of written informed consent for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
The burden of ventricular arrhythmias, defined as the total number of sustained ventricular tachycardia (sVT) events recorded during the 6-month observation period. | 6 months
  Each documented sustained ventricular tachycardia (sVT) event, captured via electrocardiogram (ECG) or intracardiac electrogram (EGM) from the CIED memory, will be subject to physician adjudication. Automatic classification of arrhythmia type, number of sVT episodes, and number of therapies performed by the CIED will be accepted only in cases where EGM recordings are unavailable, e.g., due to device memory overflow resulting from a high volume of episodes.
  sVT criteria:
  1. Meets detection criteria in the active VT or VF zone programmed in the ICD/CRT-D and triggers an appropriate therapy; or
  2. Meets detection criteria in the VT monitoring zone programmed in the ICD/CRT-D and lasts ≥ 30 seconds; or
  3. Is misclassified by the ICD/CRT-D as a supraventricular tachycardia but is reclassified as sVT after physician review of the EGM; or
  4. Is recorded on surface ECG with a duration of ≥ 30 seconds.
Absence of treatment-related serious adverse events (SAEs) during the 18-month follow-up period | 18 months
  All adverse events (AEs) assessed by the investigator as having a probable causal relationship with either the experimental therapy or standard therapy will be classified as adverse events and recorded in the study protocol.
  Serious Adverse Events (SAEs)
  Each adverse medical event meeting any of the following criteria will be classified as a Serious Adverse Event (SAE):
  * Results in the death of the patient.
  * Is life-threatening to the patient.
  * Results in permanent or significant disability or requires intervention to prevent permanent damage to tissues or organs.
  * Requires re-hospitalization or leads to an extension of the hospitalization related to the procedure by more than 24 hours.

SECONDARY OUTCOMES:
Reduction in ventricular arrhythmia burden, measured as the percentage decrease in the mean monthly number of sustained ventricular tachycardia events during the 6-month follow-up after therapy initiation, compared to corresponding period pre-treatment | 6 months
  Sustained ventricular arrhythmias will be counted as stated in the Primary Outcome Measures.
Occurrence of sVT during the 18-month follow-up period | 18 months
  Sustained ventricular arrhythmias will be counted as stated in the Primary Outcome Measures.
Time to first occurrence of sVT during the 18-month follow-up period. | 18 months
  Sustained ventricular arrhythmias will be counted as stated in the Primary Outcome Measures.
Number of appropriate ICD/CRT-D therapies delivered during the 18-month follow-up period. | 18 months
  Appropriate therapy will be defined as: a. Therapy (ATP or shock) delivered by the ICD/CRT-D due to sVT and confirmed by physician adjudication (after excluding supraventricular arrhythmias and/or sensing abnormalities); or b. External electrical or pharmacological cardioversion following physician-confirmed documentation of sVT on ECG.
  Only one therapy will be counted per sVT episode. In cases where multiple therapies are delivered sequentially during a single episode, the final effective therapy leading to episode termination will be considered and counted.
Number of hospitalizations due to arrhythmic causes during the 18-month follow-up period. | 18 months
  Number of hospitalizations due to arrhythmic causes during the 18-month follow-up period.
All-cause mortality during the 18-month follow-up period. | 18 months
  All-cause mortality during the 18-month follow-up period.
Improvement in quality of life assessed using the Polish version of the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire during the 18-month follow-up period. | 18 months
  Improvement in quality of life assessed using the Polish version of the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire during the 18-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof S. Gołba, Professor, Study Director — Department of Electrocardiology, Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University in Katowice, Ziolowa 45/47, Katowice 40-635, Poland; Danuta Łoboda, MD, PhD, Principal Investigator — Department of Electrocardiology, Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University in Katowice, Ziolowa 45/47, Katowice 40-635, Poland
Locations (1):
- Department of Electrocardiology, Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University in Katowice, Katowice, Upper-Silesia, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Due to General Data Protection Regulation (GDPR) - EU regulation on personal data protection (Regulation (EU) 2016/679).

REFERENCES:
- [Background] Miszczyk M, Sajdok M, Bednarek J, Latusek T, Wojakowski W, Tomasik B, Wita K, Jadczyk T, Kurzelowski R, Drzewiecka A, Cybulska M, Gardas R, Jarosinski G, Dolla L, Grzadziel A, Zub K, Bekman A, Kaminiow K, Kozub A, Golba KS, Blamek S. Stereotactic management of arrhythmia - radiosurgery in treatment of ventricular tachycardia (SMART-VT). Results of a prospective safety trial. Radiother Oncol. 2023 Nov;188:109857. doi: 10.1016/j.radonc.2023.109857. Epub 2023 Aug 18. PMID 37597807
- [Background] Miszczyk M, Jadczyk T, Golba K, Wojakowski W, Wita K, Bednarek J, Blamek S. Clinical Evidence behind Stereotactic Radiotherapy for the Treatment of Ventricular Tachycardia (STAR)-A Comprehensive Review. J Clin Med. 2021 Mar 17;10(6):1238. doi: 10.3390/jcm10061238. PMID 33802802
- See also: Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0, U.S. Department of Health and Human Services. Published: November 27, 2017 — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/ctcae_v5_quick_reference_5x7.pdf
- See also: NCI Guidelines For Investigators: ADVERSE EVENT REPORTING REQUIREMENTS FOR DCTD (CTEP AN D CIP) AND DCP inds AND ides — https://ctep.cancer.gov/protocoldevelopment/adverse_effects.htm
- See also: Miszczyk M, Jadczyk T, Tomasik B, et al. Stereotactic management of arrhythmia radiosurgery in treatment of ventricular tachycardia (SMART VT) clinical trial protocol and study rationale. OncoReview 2020; 10(4): 123 129. — https://www.journalsmededu.pl/index.php/OncoReview/article/view/1147